CLINICAL TRIAL: NCT04793490
Title: Efficacy and Efficiency of Sphenopalatine Ganglion Block for Management of Post-dural Puncture Headache in Obstetric Patients-A Randomized Clinical Trial
Brief Title: Sphenopalatine Ganglion Block for Management of Post- Dural Puncture Headache in Obstetric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Mostafa Mohamed Ali Mowafi, Lecturer of anesthesia ,principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R 12/2021
Record Dates: First submitted 2021-03-06; First posted 2021-03-11 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-03

CONDITIONS: Post-Dural Puncture Headache
Keywords: Sphenopalatine ganglion block; Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control group) (Other): Patients will receive paracetamol 1 g thrice daily intravenously
  Interventions: Drug: paracetamol
- Group B (Sphenopalatine ganglion block group) (Active Comparator): patients will receive sphenopalatine ganglion block via transnasal approache by a cotton tipped applicator soaked in 2%lignocaine with 4 mg dexamethasone
  Interventions: Procedure: Sphenopalatine ganglion block

INTERVENTIONS:
Procedure: Sphenopalatine ganglion block — Patients will receive the SPGB via the transnasal approache by a cotton tipped applicator soaked in lignocaine 2% with 4 mg dexamethasone
  Other Names: SPGB
  Arms: Group B (Sphenopalatine ganglion block group)
Drug: paracetamol — patients will receive paracetamol 1 g thrice daily intravenously
  Other Names: acetaminophen
  Arms: Group A (Control group)

SUMMARY:
The purpose of this trial is to study the efficacy and efficiency of sphenopalatine ganglion block for management of post dural puncture headache in obstetric patients

DETAILED DESCRIPTION:
Background and objectives: Post dural puncture headache(PDPH) is a common complication of lumbar puncture, it is likely due to the loss of cerebrospinal fluid into the epidural space through the dural tear. The prevalence of PDPH is higher in pregnant women.Sphenopalatine ganglion block (SPGB) is a non-invasive intervention with minimal adverse effects, it is indicated in acute and chronic facial/head pain like cluster headache, trigeminal neuralgia, post herpetic neuralgia and pain due to head and neck cancer.SPGB can be performed by different approaches:transnasal,transoral ,sub zygomatic and lateral infratemporal.Transnasal is the easiest, least invasive approach which can be done at bedside.

The objective of this trial is to study the efficacy and efficiency of sphenopalatine ganglion block for management of post-dural puncture headache in obstetric patients.The following will be recorded: pain score will be assessed using the numeric rating pain scale(NRS),heart rate and mean arterial pressure, onset and duration of analgesia, total dose of ketorolac, duration of hospital stay and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Female patients ASA I or II post caesarean section
* Body weight between 60-100 kg
* Active PDPH within days after spinal anesthesia not relieved with standard treatment such as, intravenous fluids, bed rest and caffeine.

Exclusion Criteria:

* Patient refusal to participate in the study
* Body mass index >35kg/m2
* Patients with :coagulopathy ,nasal septal deviation,polyp
* History of nasal bleeding
* Allergy to local anesthetic

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Numeric rating pain score | First 24 hours after the procedure
  Numeric rating pain score will be used to assess the efficacy of SPGB for treatment of PDPH

SECONDARY OUTCOMES:
Total analgesic consumption | First 24 hours after the procedure
  total dose of ketorolac will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Marwa M Mowafi, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No